CLINICAL TRIAL: NCT04160715
Title: Korean Idiopathic Pulmonary Fibrosis Registry
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jong Sun Park, Associate professor, Seoul National University Bundang Hospital
Other Study IDs: 1.1
Record Dates: First submitted 2019-10-30; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — serum, protein, DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter prospective registry of IPF patients in South Korea. The Seoul National University Bundang Hospital is the coordination center for the Korean IPF Registry built by a collaboration of the Korean Interstitial Lung Diseases (ILD) Study Group.

DETAILED DESCRIPTION:
Korean ILD Study Group includes investigators of 30 hospitals. Demographic, pulmonary function, laboratory data, chest CT findings and hospital course of IPF patients are collected.

ELIGIBILITY:
Inclusion Criteria:

* IPF patients diagnosed by multidisciplinary discussion

Exclusion Criteria:

* Other interstitial lung diseases except for IPF
* connective tissue disease-related ILD
* exposure-related ILD

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with IPF
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
survival of IPF | through study completion, an average of 1 year
  lung function change (FVC, DLCO)

SECONDARY OUTCOMES:
survival | through study completion, an average of 1 year
  death rate
acute exacerbation | through study completion, an average of 1 year
  rate of acute exacerbation
incidence of comorbidity | through study completion, an average of 1 year
  incidence of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Man Pyo Chung, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

REFERENCES:
- [Derived] Moon SW, Kim SY, Chung MP, Yoo H, Jeong SH, Kim DS, Song JW, Lee HL, Choi SM, Kim YW, Kim YH, Park CS, Park SW, Park JS, Jegal Y, Lee J, Uh ST, Kim TH, Lee JH, Kim YH, Shin B, Lee HK, Yang SH, Lee H, Kim SH, Lee EJ, Choi HS, Shin H, Park YB, Shin JW, Park MS. Longitudinal Changes in Clinical Features, Management, and Outcomes of Idiopathic Pulmonary Fibrosis. A Nationwide Cohort Study. Ann Am Thorac Soc. 2021 May;18(5):780-787. doi: 10.1513/AnnalsATS.202005-451OC. PMID 33270528